CLINICAL TRIAL: NCT05469204
Title: Effect of Gender-Affirming Estrogen Therapy on Drug Metabolism, Transport, and Gut Microbiota
Brief Title: Effect of Estrogen Treatment on Drug Metabolism and Transport
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Lauren Cirrincione, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00014091; 1K23GM147350 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Transgender Persons
Keywords: hormone therapy; estrogen treatment
MeSH Terms: interventions — Midazolam; Digoxin; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy transgender adults (Other): Healthy transgender adults will be studied on two separate study days and serve as their own control.
  Interventions: Drug: Midazolam oral solution; Drug: Digoxin Oral Tablet; Drug: Acetaminophen Oral Tablet; Drug: Midazolam Injectable Solution

INTERVENTIONS:
Drug: Midazolam oral solution — 2 mg single-dose before and during estradiol treatment.
Drug: Digoxin Oral Tablet — 0.25 mg single-dose before and during estradiol treatment.
Drug: Acetaminophen Oral Tablet — 500 mg single-dose before and during estradiol treatment.
Drug: Midazolam Injectable Solution — 1 mg intravenous single-dose before and during estradiol treatment.

SUMMARY:
This project will evaluate the effect of estrogen treatment on how other medications are processed by the body.

DETAILED DESCRIPTION:
Estradiol is prepared as a medication that patients may take to increase hormone levels. Changes in estradiol concentrations in the body may affect how the body processes other medicines. The purpose of this study is to find out how estradiol therapy affects a single tracer dose of approved medicines in the blood (midazolam, digoxin, and acetaminophen) and to confirm estradiol treatment does not affect natural bacterial in the gut.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified trans* adult 18-55 years of age.
* Not taking estradiol treatment currently.
* Planning to start injectable estradiol or estradiol tablets for gender-affirming medical care.

Exclusion Criteria:

* Unwilling/unable to return for project follow-up visits.
* Unwilling/unable to provide written informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as transgender or trans nonbinary
Enrollment: 22 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
midazolam AUC ratio (treatment/control) | 0-6 hours
  ratio of the area under of the plasma concentration time curve (AUC) of midazolam in the presence to absence of gender-affirming estradiol treatment.
digoxin renal clearance (treatment/control) | 0-48
  ratio of digoxin renal clearance in the presence to absence of gender-affirming estradiol treatment.

SECONDARY OUTCOMES:
midazolam Cmax ratio (treatment/control) | 0-6 hours
  ratio of the maximum plasma concentration (Cmax) of midazolam in the presence to absence of gender-affirming estradiol treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT05469204/ICF_000.pdf